CLINICAL TRIAL: NCT00781066
Title: Controlled Cord Traction During Third Stage of Labor: Pilot Trial
Brief Title: Controlled Cord Traction During Third Stage of Labor
Acronym: CCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad de la Republica (Other)
Collaborators: Unidad de Investigación Clínica y Epidemiológica Montevideo (Other); Institute for Clinical Effectiveness and Health Policy (Other)
Responsible Party: Alicia Aleman, Clinical and Epidemiological Research Unit Montevideo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCT 06-00051; D43TW005492 (NIH grant number); D43TW005492 (NIH)
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2008-10-28 (Estimated); Status verified 2008-10

CONDITIONS: Postpartum Hemorrhage
Keywords: POSTPARTUM HEMORRHAGE; PREVENTION; CORD TRACTION; THIRD STAGE LABOR
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Controlled cord traction (CCT)
  Interventions: Procedure: Controlled cord traction
- 2 (Active Comparator): No CCT
  Interventions: Procedure: No controlled cord traction

INTERVENTIONS:
Procedure: Controlled cord traction — 1. Clamp the cord close to the perineum (once pulsation stops, or after three minutes in a healthy newborn), hold it in one hand.
  2. Place the other hand just above the woman's pubic bone and stabilize the uterus by applying counter-pressure during controlled cord traction.
  3. Keep slight tension on the cord and await a strong uterine contraction (2-3 minutes).
  4. With the strong uterine contraction, encourage the mother to push and very gently pull downward on the cord to deliver the placenta. Continue to apply counter-pressure to the uterus.
  5. If the placenta does not descend during 30-40 seconds of CCT, do not continue to pull on the cord:
     * Gently hold the cord and wait until the uterus is well contracted again;
     * With the next contraction, repeat CCT with counter-pressure.
  Arms: 1
Procedure: No controlled cord traction — 1. Clamp the cord close to the perineum (once pulsation stops, or after three minutes in a healthy newborn).
  2. No CCT will be used and no fundal pressure. The placenta will be delivered physiologically, and signs for placental separation will be awaited (gush of blood from the vagina, descent of the umbilical cord, and increase in the height of the uterus in the abdomen as the lower segment was distended).
  3. After separation, delivery of the placenta will be aided only by maternal expulsive efforts and/or gravity.
  Arms: 2

SUMMARY:
Of the estimated number of 529,000 maternal deaths for the year 2000, 132,000 (25%) were caused by postpartum hemorrhage (PPH); 99% of these deaths occurred in low-income countries. Where maternal mortality is high and resources are limited, the introduction of low-cost, evidence-based practices for primary prevention of PPH is an urgent need. Controlled cord traction (CCT) is actively promoted in combination with prophylactic uterotonics for the prevention of PPH. While the administration of uterotonics has been proven effective, there is no evidence of CCT being beneficial or safe. The investigators propose this study to evaluate two primary questions:

1. In women having term, single vaginal deliveries in hospital settings, in whom the third stage is managed with prophylactic oxytocin, does CCT produce a clinically significant reduction in the incidence of postpartum blood lose?
2. In these women, does CCT produce a clinically significant increase in the incidence of severe complications, including uterine inversion or the need for subsequent surgical evacuation of retained placental tissues and membranes (curettage or manual removal)?

To answer these two questions we designed two arms randomized controlled trial.

DETAILED DESCRIPTION:
Subjects This study will be conducted in two Public Hospital from Montevideo, Uruguay. A total of 200 women (100 by group) will be recruited.

Description of the Study Design This will be a two-arm, randomized controlled clinical trial in which 200 women having a single vaginal delivery and receiving prophylactic oxytocin for the management of the third stage of labor at two public hospital in Montevideo will be allocated to one of two interventions: CCT or a "hands-off" policy. All outcomes will be measured before maternal discharge from the hospital. The primary outcome is postpartum blood loss.

Duration of the Study We estimate that we will need a total of 11 months to complete this study. Three months will be needed for preparation (installing data collection resources and training data collectors and birth attendants), and 6 months for recruitment, and two months for data analysis and preparation of reports and manuscripts.

Where Subjects Are/ Study Site and Populations The study will be conducted in two public hospitals from Montevideo, Uruguay. These are third level public hospitals supported by the University of the Republic, with a total of 9,900 deliveries per year.

Full Description of Risks There is no evidence to suggest that there were risks from this study to the women or the newborns, because it is not known if CCT is associated with serious complications in the mother. In all previous active management trials and in the two CCT trials, there were no reported cases of uterine inversion, and currently, CCT is the recommended standard of care during delivery. In theory, the most severe potential complication is uterine inversion, which can be a life-threatening condition if adequate care is not provided. However, this event is unlikely with the simultaneous use of uterotonics to assure a well contracted uterus and eventually, it can be successfully managed in hospital settings.

Benefits for Subjects and/or Society:

We do not expect a clinical and important benefit from this study at an individual level of the pregnant women. However, this study will provide useful information to evaluate one specific intervention recommended for the management of third stage of labor.

Inducement for Participants:

No monetary inducement will be offered to the participants.

Costs to Subjects: N/A

Statistical Analysis Before addressing the research question, descriptive statistics and summary graphics such as histograms will be prepared and examined for outcomes and demographic variables. All analyses addressing the study research questions will use the "intention to treat" principle, thus comparing the original intervention group to the original nonintervention group, even if individuals have withdrawn from the study or shifted to another group. The analysis plan and presentation of results will follow the recommendation of the CONSORT statement. In this study the primary outcome is continues (blood loss), therefore, median and inter-quartile ranges will be computed as part of descriptive data analysis to understand the distribution of the outcome variables and to assess the need of data transformation or adoption of nonparametric tests, including Mann-Whitney U tests. Means for the two groups will be compared by the two-sample t-test. A similar analysis will be performed for the duration (in minutes) of the third stage of labor.

Methods of Recruitment:

Enrollment will be done during and previous to women's labor at the maternity. Screening will start at the time of admission and when possible during prenatal care, and for those eligible women, a signed consent form will be required. Sealed envelopes opened just before delivery(at delivery guard) will be used to determine whether the woman should receive CCT or not. A random allocation scheme will be derived from a computer-generated list of numbers, with randomly permuted blocks.

Informed Consent Services directors will provide written authorization to participate in this study. Individual birth attendants will receive an information sheet describing the objectives of the study and including the name and phone number of the study coordinator. Birth attendants will also be invited to participate in the training workshops. Women will be invited to participate upon admission to the hospital (or during prenatal care when possible) and, if they agree to participate, will provide written informed consent to their birth attendant. The birth attendant will then be required to disclose to the patient all of the facts about the nature of the trial, interventions under comparison, the risks involved, available alternatives and their risk, and reasonable expectations for the treatment outcome. This study was submitted to the Institutional Review Board of the School of Medicine, University of Uruguay for approval and the Institutional Review Board of Tulane University . The PI and co-PI have attended training sessions on the protection of human subjects and have been certified by the Institutional Review Boards at their institutions. The coordinator and research assistant invited to participate in this study will be asked to complete an on-line training session on protection of human subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or more
* Single pregnant women during third trimester of prenatal care or in early first stage of labor at the participating hospital (Cervical dilatation ≤ 6 cm).
* No indication of cesarean section
* No contraindications for receiving prophylactic uterotonics
* Gestational age ≥ 37 weeks

Additional Inclusion Criteria for Randomization

* Imminent vaginal delivery

Exclusion Criteria:

* Severe acute complications during labor requiring emergency actions (e.g., eclampsia, hemorrhage, or any other complications that imply serious difficulties according to the judgment of the attendant)
* No consent to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Postpartum blood loss | a minimum of 20 minutes after delivery

SECONDARY OUTCOMES:
Manual removal of placenta | within 1 hour after delivery
Uterine inversion | within 30 minutes after delivery
Uterine curettage | before hospital discharge
Blood transfusion | before Hospital discharge
Length of third stage of labor (minutes) | until expulsion of the placenta

CONTACTS AND LOCATIONS:
Overall Officials: Alicia V Aleman, MD, Principal Investigator — Unidad de Investigación Clínica y Epidemiológica Montevideo
Locations (2):
- Uruguay (2):
  - Clinica's Hospital Manuel Quintela of the University of the Republic of Uruguay, Montevideo, Montevideo Department
  - Pereira Rossell Hospital, Montevideo, Montevideo Department

REFERENCES:
- [Derived] Carvalho JF, Piaggio G, Wojdyla D, Widmer M, Gulmezoglu AM. Distribution of postpartum blood loss: modeling, estimation and application to clinical trials. Reprod Health. 2018 Dec 4;15(1):199. doi: 10.1186/s12978-018-0641-1. PMID 30514326
- [Derived] Piaggio G, Carvalho JF, Althabe F. Prevention of postpartum haemorrhage: a distributional approach for analysis. Reprod Health. 2018 Jun 22;15(Suppl 1):97. doi: 10.1186/s12978-018-0530-7. PMID 29945633
- See also: School of Medicine of the University of the Republic — http://www.fmed.edu.uy/
- See also: Clinical and Epidemiological Research Unit Montevideo — http://www.unicem-web.org/